CLINICAL TRIAL: NCT05324124
Title: An Open-Label, Randomized, Two-Period Crossover Study to Investigate the Effect of Food on the Pharmacokinetics of Selpercatinib in Healthy Participants
Brief Title: A Study of the Effect of Food on Selpercatinib (LY3527723) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Loxo Oncology, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18178; J2G-MC-JZPA (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: Selpercatinib; Food; Pharmacokinetics
MeSH Terms: interventions — selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Selpercatinib (Fasted/Fed) (Experimental): Period 1: 160 milligrams (mg) Selpercatinib administered orally on Day 1 in fasted state.
  Period 2: 160 mg Selpercatinib administered orally on Day 8 in fed state.
  Interventions: Drug: Selpercatinib
- Selpercatinib (Fed/Fasted) (Experimental): Period 1: 160 mg Selpercatinib administered orally on Day 1 in fed state.
  Period 2: 160 mg Selpercatinib administered orally on Day 8 in fasted state.
  Interventions: Drug: Selpercatinib

INTERVENTIONS:
Drug: Selpercatinib — Administered orally.
  Other Names: LY3527723; LOXO-292

SUMMARY:
The main purpose of this study is to learn about how food affects selpercatinib in healthy participants. The selpercatinib will be administered in fed and fasted states. Participation could last about 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, vital signs and clinical laboratory tests.

Exclusion Criteria:

* Have a history or presence of cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Selpercatinib Fasted/Fed: 160 milligrams (mg) Selpercatinib will be administered orally on Day 1 in fasted state and on Day 8 in fed state.
- Selpercatinib Fed/Fasted: 160 mg Selpercatinib will be administered orally on Day 1 in fed state and on Day 8 in fasted state.
Period: Period 1
Arm/Group | Selpercatinib Fasted/Fed | Selpercatinib Fed/Fasted
Started | 23 | 23
Received One Dose of Study Drug | 23 | 23
Completed | 22 | 22
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1
Period: Period 2
Arm/Group | Selpercatinib Fasted/Fed | Selpercatinib Fed/Fasted
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Selpercatinib: 160 mg Selpercatinib will be administered orally on Day 1 in fasted state or fed state and on Day 8 in fed state or fasted state.
Arm/Group | Selpercatinib
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 45
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 46

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics(PK): Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Selpercatinib
Description: PK: AUC[0-∞] of Selpercatinib'
Time Frame: PK: Day 1 and Day 8: Predose, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, and 72 hours (h) postdose;
Population: All participants who received doses of study drug on Day 1 and Day 8 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram * hour per milliliter (ng*hr/mL
Groups:
- Selpercatinib Fasted (Reference): 160 mg Selpercatinib administered orally in fasted state.
- Selpercatinib Fed (Test): 160 mg Selpercatinib administered orally in fed state.
Arm/Group | Selpercatinib Fasted (Reference) | Selpercatinib Fed (Test)
Number analyzed (Participants) | 44 | 44
nanogram * hour per milliliter (ng*hr/mL | 23400 (32) | 22500 (44)
Statistical Analysis 1: Comparison: Selpercatinib Fasted (Reference) vs Selpercatinib Fed (Test); Test type: Other; Ratio of Geometric Least Squares Mean = 0.952, 90% CI 2-sided [0.876 to 1.03]

2. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Measured Concentration Value (AUC[0-tlast]) of Selpercatinib
Description: PK: AUC[0-tlast] of Selpercatinib
Time Frame: PK: Day 1 and Day 8: Predose, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, and 72 hours (h) postdose;
Population: All participants who received doses of study drug on Day 1 and Day 8 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Selpercatinib Fasted (Reference) | Selpercatinib Fed (Test)
Number analyzed (Participants) | 44 | 44
ng*hr/mL | 22700 (32) | 21700 (46)
Statistical Analysis 1: Comparison: Selpercatinib Fasted (Reference) vs Selpercatinib Fed (Test); Test type: Other; Ratio of Geometric Least Squares Mean = 0.949, 90% CI 2-sided [0.869 to 1.04]

3. Primary Outcome: PK: Maximum Concentration (Cmax) of Selpercatinib
Description: PK: Cmax of Selpercatinib.
Time Frame: PK: Day 1 and Day 8: Predose, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, and 72 hours (h) postdose;
Population: All participants who received doses of study drug on Day 1 and Day 8 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Selpercatinib Fasted (Reference) | Selpercatinib Fed (Test)
Number analyzed (Participants) | 44 | 44
nanograms per milliliter (ng/mL) | 1840 (39) | 1540 (45)
Statistical Analysis 1: Comparison: Selpercatinib Fasted (Reference) vs Selpercatinib Fed (Test); Test type: Other; Ratio of Geometric Least Squares Mean = 0.829, 90% CI 2-sided [0.744 to 0.925]

ADVERSE EVENTS:
Time Frame: Screening up to 21 days
Description: All participants who received at least one dose of study drug.
Groups:
- 160 mg Selpercatinib Fasted: 160 milligrams (mg) Selpercatinib will be administered orally on Day 1 in fasted state and on Day 8 in fed state.
- 160 mg Selpercatinib Fed: 160 mg Selpercatinib will be administered orally on Day 1 in fed state and on Day 8 in fasted state.
Arm/Group | 160 mg Selpercatinib Fasted | 160 mg Selpercatinib Fed
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 29/45 | 21/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 160 mg Selpercatinib Fasted (N=45) | 160 mg Selpercatinib Fed (N=45)
Diarrhoea (Gastrointestinal disorders) | 7 (11) | 5 (13)
Catheter site bruise (General disorders) | 7 (7) | 4 (4)
Catheter site erythema (General disorders) | 12 (12) | 13 (14)
Catheter site pain (General disorders) | 10 (13) | 6 (8)
Catheter site swelling (General disorders) | 3 (7) | 3 (3)
Fatigue (General disorders) | 4 (4) | 3 (3)
Vessel puncture site bruise (General disorders) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 6 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT05324124/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT05324124/SAP_001.pdf